CLINICAL TRIAL: NCT06222164
Title: The Use of Residual De-identified Specimens and/or Samples From Patients for Clinical Research
Status: Recruiting | Type: Observational
Sponsor: Invivoscribe, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IVS-010-003
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Hematologic Diseases
Keywords: residual samples hematologic diseases
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual specimen/sample collection study where peripheral blood (PB), bone marrow (BM), genomic (gDNA), and/or formalin-fixed paraffin-embedded tissue (FFPE) specimens/samples are obtained from patient samples sent to LabPMM, LLC for clinical testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Residual Specimens: Residual specimen/sample collection study where peripheral blood (PB), bone marrow (BM), genomic (gDNA), and/or formalin-fixed paraffin-embedded tissue (FFPE) specimens/samples are obtained from patient samples sent to LabPMM, LLC for clinical testing.

SUMMARY:
Acquire residual human specimens and/or samples from patient samples which were sent for testing at LabPMM, LLC for Clinical Research

DETAILED DESCRIPTION:
Residual specimen/sample collection study where peripheral blood (PB), bone marrow (BM), genomic (gDNA), and/or formalin-fixed paraffin-embedded tissue (FFPE) specimens/samples are obtained from patient samples sent to LabPMM, LLC for clinical testing. Samples may be used for Clinical Research at LabPMM, LLC or at partner institutions

ELIGIBILITY:
Inclusion Criteria:

1. Specimen/sample, peripheral blood (PB), bone marrow (BM), genomic DNA (gDNA) and/or formalin-fixed paraffin-embedded tissue (FFPE) from patients whose specimens/samples have been sent to LabPMM for clinical testing
2. Donor Age ≥ 18 years

Exclusion Criteria:

1. Sample/specimen has been obtained from a third-party vendor with a Materials Transfer Agreement (MTA) on file with LabPMM
2. The specimens/samples have previously been enrolled in a clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Specimen/sample, peripheral blood (PB), bone marrow (BM), genomic DNA (gDNA) and/or formalin-fixed paraffin-embedded tissue (FFPE) from patients whose specimens/samples have been sent to LabPMM for clinical testing
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-03-30 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Enrollment | 3 years
  N=2000

CONTACTS AND LOCATIONS:
Locations (1):
- LabPMM, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Study uses residual de-identified human samples

REFERENCES:
- See also: Related Info — https://invivoscribe.com